CLINICAL TRIAL: NCT06262360
Title: Changes in Pulmonary Ventilation Distribution Assessed by EIT (Electrical Impedance Tomography) in Healthy Children Under General Anesthesia; a Pilot Study Comparing Mask Spontaneous Breathing and Laryngeal Mask Spontaneous Breathing With and Without Ventilatory Support
Brief Title: Changes in Pulmonary Ventilation Distribution Assessed by Electrical Impedance Tomography in Healthy Children Under General Anesthesia
Acronym: EIT_ped
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: P2023457
Record Dates: First submitted 2024-02-06; First posted 2024-02-16 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia, Pediatric
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia with spontaneous mask ventilation (Experimental): Patients under general anesthesia with spontaneous mask ventilation
  Interventions: Procedure: General anesthesia with mask ventilation
- General anesthesia and spontaneous laryngeal mask ventilation (Experimental): Patients under general anesthesia and spontaneous laryngeal mask ventilation
  Interventions: Procedure: General anesthesia and spontaneous laryngeal mask ventilation
- General anesthesia with spontaneous laryngeal mask ventilation with pressure support (Experimental): Patients under general anesthesia with spontaneous laryngeal mask ventilation with pressure support
  Interventions: Procedure: General anesthesia with spontaneous laryngeal mask ventilation with pressure support

INTERVENTIONS:
Procedure: General anesthesia with mask ventilation — Randomization to General anesthesia with mask ventilation
  Arms: General anesthesia with spontaneous mask ventilation
Procedure: General anesthesia and spontaneous laryngeal mask ventilation — Randomization to General anesthesia and spontaneous laryngeal mask ventilation
  Arms: General anesthesia and spontaneous laryngeal mask ventilation
Procedure: General anesthesia with spontaneous laryngeal mask ventilation with pressure support — Randomization to General anesthesia with spontaneous laryngeal mask ventilation with pressure support
  Arms: General anesthesia with spontaneous laryngeal mask ventilation with pressure support

SUMMARY:
The incidence of atelectasis is high in patients undergoing general anesthesia. This may cause oxygenation impairment and further contribute to post-operative pulmonary complications. As important airway management devices for general anesthesia, few studies have compared the impact of laryngeal mask airway and spontaneous breathing on atelectasis. Through the study, the distribution of the pulmonary ventilation of children undergoing an elective and standard procedure in our center (H.U.D.E.R.F.) will be studied using electric impedance tomography.

Children from 1 year-old to 6-year-old, ASA physical status I or II who will undergo elective circumcisions under general anesthesia associated with regional anesthesia (Penile Block10) at the One Day Clinic of H.U.D.E.R.F. (Hôpital des Enfants Reine Fabiola - Brussels - Belgium).

Patients will be allocated to three different group in a ration of 1:1:1.

* Group 1: spontaneous mask ventilation (20 patients).
* Group 2: spontaneous laryngeal mask (LMA) ventilation (20 patients).
* Group 3: spontaneous-pressure support LMA ventilation (LMA SV-PS) (20 patients).
* Standard monitoring for the inductions of the anesthesia will include non-invasive blood pressure (NIBP), pulse oximetry (SpO2), Electrocardiogram (ECG), End-Tidal CO2 (EtCO2), End Tidal Sevoflurane concentration (EtSev %), inspired fraction of oxygen (FiO2), body temperature (rectal thermometer).

Induction is based as well on the local routine protocols using an inhalation induction of the patient with Sevoflurane (Fet of 6-8%) and a recommended FiO2 from 80-90% maximum until the stabilization of the induction. Then the FiO2 will be decreased at least under 40% and Sevoflurane adapted to the need of the deepness of the anesthesia (both at the discretion of the anesthesiologist in charge of the patient).

Depending on the randomization, the patient will undergo the surgery either with spontaneous face mask ventilation (group 1), LMA spontaneous ventilation (group 2), or LMA SV-PS (group 3) (during which the pressure support will be adapted at the discretion of the anesthesiologist but with a tidal volume included in the range of 6-10ml/kg).

Electrical impedance tomography measurements:

The effects of the spontaneous breathing (mask ventilation or LMA) or the pressure support ventilation (LMA SV-PS) on atelectasis formations and the distribution of the ventilation will be assessed using electrical impedance tomography.

The device used during the study will be the "PulmoVista 500"; it will be provided by Dräger (Lübeck, Germany) free of charge and without any obligation or results/conclusions requested by Dräger. The device is approved CE (European regulation) and will be used in the conditions for which it has been designed.

A reusable belt with 16 evenly spaced electrodes will be placed around the chest of each patient included in the study between the 4th and 6th ribs as recommended by Dräger.

The EIT measurements will be taken of 4 different moments:

T1: Before induction of the anesthesia in the preoperatory waiting room (and at least 30 min after the premedication).

T2: After the induction of anesthesia (GA and penile block), just before the beginning of the surgical procedure.

T3: After the end of the surgical procedure, just before discontinuing the general anesthesia.

T4: Before the discharge of the PACU.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing elective circumcision
* Age 1 to 6 years
* ASA class I or II

Exclusion Criteria:

* Any history of lung diseases, congenital heart diseases or abdominal diseases that could interfere with lungs dynamic.
* ASA physical status11 > II.
* Patients whose weight is less than 10 kg.
* The use of Jackson-Rees device12.
* Contraindication for premedication.
* Contraindication for mask ventilation or laryngeal mask ventilation13.
* Contraindication for regional anesthesia.
* Need for opioids administration during surgery.
* Patients with uncontrollable movements of the body.
* Inability of parents/tutors to understand French or Dutch.
* Patients whose parents do not agree with their participation in the study
* Patients with thoracic perimeters (between 4th and 6th ribs) less than 37.5 cm (minimal size for the pediatric EIT belt) or more than 72 cm (maximal size for the pediatric EIT belt)
* Patients with damaged skin or impaired skin contact of the electrodes due to wound dressings.
* Patients with spinal lesions or fractures (acute or recent)
* Patients with pacemaker, defibrillators, or other electrically active implants

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Variation of poorly ventilated pulmonary zones | 4 hours
  Primary outcome will be the variation of poorly ventilated zones between period T1 (before induction of anesthesia) and period T2 (at the discharge from the PACU) that we may surrogate as atelectasis. The Pulmovista device divides the lungs in 4 areas (front to back in a supine patient) and the percentage of ventilation going to each area is measure by electric impedance variation. The difference in the distribution between the 4 areas will be measured (expressed as % of total ventilation).

CONTACTS AND LOCATIONS:
Locations (1):
- H.U.B - Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nascimento MS, Rebello CM, Costa ELV, Correa LC, Alcala GC, Rossi FS, Morais CCA, Laurenti E, Camara MC, Iasi M, Apezzato MLP, do Prado C, Amato MBP. Effect of general anesthesia and controlled mechanical ventilation on pulmonary ventilation distribution assessed by electrical impedance tomography in healthy children. PLoS One. 2023 Mar 16;18(3):e0283039. doi: 10.1371/journal.pone.0283039. eCollection 2023. PMID 36928465
- [Background] Clasen D, Winter I, Rietzler S, Wolf GK. Changes in ventilation distribution during general anesthesia measured with EIT in mechanically ventilated small children. BMC Anesthesiol. 2023 Apr 12;23(1):118. doi: 10.1186/s12871-023-02079-z. PMID 37046213
- [Background] Ji SH, Jang HS, Jang YE, Kim EH, Lee JH, Kim JT, Kim HS. Effect of spontaneous breathing on atelectasis during induction of general anaesthesia in infants: A prospective randomised controlled trial. Eur J Anaesthesiol. 2020 Dec;37(12):1150-1156. doi: 10.1097/EJA.0000000000001327. PMID 33009186
- [Background] Durlak W, Kwinta P. Role of electrical impedance tomography in clinical practice in pediatric respiratory medicine. ISRN Pediatr. 2013 Dec 25;2013:529038. doi: 10.1155/2013/529038. eCollection 2013 Dec 25. PMID 24455294
- [Background] Li X, Liu B, Wang Y, Xiong W, Zhang Y, Bao D, Liang Y, Li L, Liu G, Jin X. The effects of laryngeal mask airway versus endotracheal tube on atelectasis in patients undergoing general anesthesia assessed by lung ultrasound: A protocol for a prospective, randomized controlled trial. PLoS One. 2022 Sep 9;17(9):e0273410. doi: 10.1371/journal.pone.0273410. eCollection 2022. PMID 36084154
- [Background] Riva T, Pascolo F, Huber M, Theiler L, Greif R, Disma N, Fuchs A, Berger-Estilita J, Riedel T. Evaluation of atelectasis using electrical impedance tomography during procedural deep sedation for MRI in small children: A prospective observational trial. J Clin Anesth. 2022 May;77:110626. doi: 10.1016/j.jclinane.2021.110626. Epub 2021 Dec 10. PMID 34902800
- [Background] Froessler B, Brommundt J, Anton J, Khanduja R, Kuhlen R, Rossaint R, Coburn M. Spontaneously breathing anesthetized patients with a laryngeal mask airway: positive end-expiratory pressure does not improve oxygen saturation. Anaesthesist. 2010 Nov;59(11):1003-4, 1006-7. doi: 10.1007/s00101-010-1764-0. Epub 2010 Sep 11. PMID 20835692
- [Background] Trachsel D, Svendsen J, Erb TO, von Ungern-Sternberg BS. Effects of anaesthesia on paediatric lung function. Br J Anaesth. 2016 Aug;117(2):151-63. doi: 10.1093/bja/aew173. PMID 27440626
- [Background] Humphreys S, Pham TM, Stocker C, Schibler A. The effect of induction of anesthesia and intubation on end-expiratory lung level and regional ventilation distribution in cardiac children. Paediatr Anaesth. 2011 Aug;21(8):887-93. doi: 10.1111/j.1460-9592.2011.03547.x. Epub 2011 Mar 14. PMID 21395895
- [Background] Nascimento MS, Rebello CM, Costa ELV, Rossi FS, do Prado C, Amato MBP. Pulmonary Aeration and Posterior Collapse Assessed by Electrical Impedance Tomography in Healthy Children: Contribution of Anesthesia and Controlled Mechanical Ventilation. Anesthesiology. 2022 Nov 1;137(5):648-650. doi: 10.1097/ALN.0000000000004321. No abstract available. PMID 35930425
- [Background] Spinelli E, Mauri T, Fogagnolo A, Scaramuzzo G, Rundo A, Grieco DL, Grasselli G, Volta CA, Spadaro S. Electrical impedance tomography in perioperative medicine: careful respiratory monitoring for tailored interventions. BMC Anesthesiol. 2019 Aug 7;19(1):140. doi: 10.1186/s12871-019-0814-7. PMID 31390977
- [Background] Radke OC, Schneider T, Heller AR, Koch T. Spontaneous breathing during general anesthesia prevents the ventral redistribution of ventilation as detected by electrical impedance tomography: a randomized trial. Anesthesiology. 2012 Jun;116(6):1227-34. doi: 10.1097/ALN.0b013e318256ee08. PMID 22531334
- [Background] Hochhausen N, Kapell T, Durbaum M, Follmann A, Rossaint R, Czaplik M. Monitoring postoperative lung recovery using electrical impedance tomography in post anesthesia care unit: an observational study. J Clin Monit Comput. 2022 Aug;36(4):1205-1212. doi: 10.1007/s10877-021-00754-5. Epub 2021 Sep 20. PMID 34542735
- [Background] Wang Y, Xu H, Li H, Cheng B, Fang X. Lung aeration and ventilation after general anesthesia in left lateral position: a prospective observational study using electrical impedance tomography. Ann Palliat Med. 2021 Feb;10(2):1285-1295. doi: 10.21037/apm-20-1029. Epub 2020 Oct 9. PMID 33040550
- [Background] Brabant O, Crivellari B, Hosgood G, Raisis A, Waldmann AD, Auer U, Adler A, Smart L, Laurence M, Mosing M. Effects of PEEP on the relationship between tidal volume and total impedance change measured via electrical impedance tomography (EIT). J Clin Monit Comput. 2022 Apr;36(2):325-334. doi: 10.1007/s10877-021-00651-x. Epub 2021 Jan 25. PMID 33492490